CLINICAL TRIAL: NCT07104435
Title: A Community-Based Recreation Program to Improve Function and Quality of Life in Older Adults
Brief Title: Community Recreation to Enhance Function in Aging
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Nikhil Satchidanand, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1193595
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Physical Functional Impairment; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exergaming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No artmaking, no exergaming
- Artmaking and Exergaming (Experimental): Weekly group-based visual artmaking and dual-task exergaming
  Interventions: Other: Artmaking and exergaming

INTERVENTIONS:
Other: Artmaking and exergaming — Weekly visual artmaking and exergaming
  Arms: Artmaking and Exergaming

SUMMARY:
This aim of this study is to examine the therapeutic impacts of a group-based recreational program that delivers guided visual artmaking and dual-task exergaming, to older adults. Outcomes of interest include cognitive function (attention, task-switching, interference inhibition), physical function (balance, walking, lower-limb strength), and dual-task performance. Key implementation outcomes including intervention fidelity, feasibility, and acceptability will be explored to inform design of future community-based intervention programs.

ELIGIBILITY:
Inclusion Criteria:

* Have no more than MCI (Montreal Cognitive Assessment score ≥ 24 points)
* Have no contraindications to exercise guided by the American College of Sports Medicine (ACSM)
* Fluent in English

Exclusion Criteria:

* Have a condition that would prevent safe participation in the exercise, as determined by the Physical Activity Readiness Questionnaire for Older Adults
* Have severe neurological disease.
* Have severe psychiatric illness.
* Have a likelihood of withdrawing from the study due to severe illness or a life expectancy of < 6 mo.
* Having a lower or upper limb amputation

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-05-11 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in performance on the Stroop Color-Word Test | From enrollment to study end at 24 weeks
  Change in score on the Stroop Color-Word Test
Performance on the Trail Making Test | From baseline to study end at 24 weeks
  Change in score on the Trail Making Test

SECONDARY OUTCOMES:
Performance on Four Stage Balance Test | From baseline to study end at 24 weeks
  Change in score on the Four Stage Balance Test
Performance on the Six-Minute Walk Test | From baseline to study end at 24 weeks
  Change in score on the Six-Minute Walk Test
Dual-Task Ability | From baseline to study end at 24 weeks
  Change in scores on the Timed Up and Go Test: Dual Task

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, Buffalo, New York, United States